CLINICAL TRIAL: NCT02314754
Title: Outpatient Medical Abortion With Mifepristone and Misoprostol Through 77 Days of Gestation: A Non-inferiority Trial
Brief Title: Outpatient Medical Abortion With Mifepristone and Misoprostol Through 77 Days of Gestation
Acronym: XXGA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Gynuity Health Projects (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 1016
Record Dates: First submitted 2014-12-04; First posted 2014-12-11 (Estimated); Last update posted 2016-07-14 (Estimated); Status verified 2016-07

CONDITIONS: Medical Abortion

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 71-77 days gestational age (Experimental): Women whose pregnancies are estimated to have a gestational age of 71-77 days.
  Interventions: Drug: Mifepristone followed by misoprostol 24-48 hours later
- 64-70 days gestational age (No Intervention): Women whose pregnancies are estimated to have a gestational age of 64-70 days.( Women in this arm receive the standard of care for medical termination of pregnancy in the stated gestational age range).

INTERVENTIONS:
Drug: Mifepristone followed by misoprostol 24-48 hours later — 200mg oral mifepristone and 800mcg buccal misoprostol 24-48 hours after mifepristone
  Arms: 71-77 days gestational age

SUMMARY:
To demonstrate non-inferiority of the efficacy of 200 mg mifepristone followed in 24 to 48 hours by 800 µg buccal misoprostol in outpatient medical abortion services among women 71-77 days' compared to women 64-70 days' LMP.

ELIGIBILITY:
Inclusion Criteria:

* intrauterine pregnancy between 64 days and 77 days' LMP
* eligible for medical abortion according to study doctor assessment
* willing and able to sign consent form
* speak english or spanish (in US sites); speak the local language(s) (in international sites)
* agree to comply with the study procedures and visit schedule

Exclusion Criteria:

* Have known allergies or present other contraindications to mifepristone or misoprostol

Ages: 11 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 719 (Actual)
Dates: Start 2014-12; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Efficacy as determined by the proportion of successful terminations without surgical intervention (suction curettage or D&C) for any reason | 7-36 days
  Efficacy of medical abortion in the later first trimester as determined by the proportion of successful terminations without surgical intervention (suction curettage or D&C) for any reason

SECONDARY OUTCOMES:
Proportion of Individual Side Effects Experienced by Participants | 7-14 days
  Side effects include diarrhea, nausea, vomiting, fever, chills, headaches, dizziness and/or weakness experienced by participants
Proportion of Women Who Determine Method Acceptable | 7-14 days
  overall acceptability, time to complete abortion, bleeding, side effects, pain
Proportion of Providers Who Determine Method Acceptable | 7-36 days
  As assessed by service provider semi-structured interviews

CONTACTS AND LOCATIONS:
Overall Officials: Beverly Winikoff, MD,MPH, Principal Investigator — Gynuity Health Projects
Locations (8):
- United States (4):
  - Hartford GYN Center, Hartford, Connecticut
  - Atlanta Women's Center, Atlanta, Georgia
  - John H. Stroger, Jr. Hospital of Cook CountY, Chicago, Illinois
  - Family Planning Associates Medical Group, Chicago, Illinois
- Scientific Research Institute of Obstetrics and Gynecology, Baku, Azerbaijan
- David Gagua Clinic, Tbilisi, Georgia
- Clínica Comunitaria Santa Catarina, Mexico City, Mexico
- Hung Vuong Hospital, Ho Chi Minh City, Vietnam